CLINICAL TRIAL: NCT05720559
Title: Early Blocking Strategy for Metachronous Liver Metastasis of Colorectal Cancer Based on Pre-hepatic CTC Detection
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230201zzg
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Preventive Effect of Quintuple Therapy on Metachronous Liver Metastases in Patients With Colorectal Cancer
MeSH Terms: interventions — Oxaliplatin; S 1 (combination); Cetuximab; Metronidazole; Vitamin A; Folic Acid; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment group (Experimental): Conventional treatment was performed according to the NCCN Guidelines for Colorectal Cancer 2023 Edition
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine
- Quintuple method treatment group (Experimental): SOX regimen chemotherapy, low dose cetuximab targeted therapy, and folic acid, vitamin A, metronidazole three-drug regimen were combined. Specific drug dosages were as follows: SOX regimen was administered every three weeks, d1 was given oxaliplatin intravenously, the dosage was 130mg/ m2 * patient's body surface area, d2-d15 was taken orally by S1, 20mg three times a day each time. Cetuximab combined with chemotherapy was administered intravenously, once every three weeks, before oxaliplatin, and the dosage was 250mg/ m2 * patient's body surface area. Metronidazole 0.4g/ time, once a day; Vitamin A 25,000 units/time, once a day; Folic acid 0.4mg/ time, once a day. The last three drugs were continued until the end of all chemotherapy cycles. These regimens last for 6 to 8 sessions.
  Interventions: Drug: Oxaliplatin; Drug: S1; Drug: Cetuximab; Drug: Metronidazole; Drug: Vitamin A; Drug: Folic acid

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin via intravenous drip on d1 at a dose of 130mg/m2 × patient 's body surface area
Drug: S1 — Orally on d2-d15 at 20 mg three times daily
  Arms: Quintuple method treatment group
Drug: Cetuximab — Cetuximab combined with chemotherapy was administered simultaneously, once every three weeks,and intravenous drip was performed before oxaliplatin at a dose of 250 mg/m2 × body surface area.
  Arms: Quintuple method treatment group
Drug: Metronidazole — Metronidazole 0.4g/time, qd
  Arms: Quintuple method treatment group
Drug: Vitamin A — Vitamin A 25,000 units/time, qd
  Arms: Quintuple method treatment group
Drug: Folic acid — Folic acid 0.4 mg/time, qd
  Arms: Quintuple method treatment group
Drug: Capecitabine — Capecitabine via orally on d2-d15 two times daily at a dose of 1000mg/m2 × patient 's body surface area.
  Arms: Conventional treatment group

SUMMARY:
In this study, the Quintuple method was applied for early intervention of prehepatic CTC-positive bowel cancer patients without dominant liver metastasis, aiming to explore the blocking effect of the Quintuple method on the metachronous liver metastases of colorectal cancer. A one-arm randomized clinical trial was conducted, and the patients were grouped according to their treatment methods. The patients with metachronous liver metastases were used as the end point of the experiment to evaluate the blocking effect of quintuple therapy.

DETAILED DESCRIPTION:
Patients diagnosed with colorectal cancer, clinical stage I to III, underwent radical surgery, and prehepatic CTC≥1 were enrolled. Patients were randomly divided into Conventional treatment group and Quintuple method treatment group. Patients in the Conventional treatment group received conventional treatment according to the NCCN Guidelines for Colorectal Cancer 2023 edition. For patients in the Quintuple method treatment group, Quintuple method intervention was adopted, that is, combined with SOX regimen chemotherapy, low-dose cetuximab targeted therapy and three-drug regimen of folic acid, vitamin A and metronidazole. Specific drug dosages were as follows: SOX regimen was administered every three weeks, d1 was given oxaliplatin intravenously, the dosage was 130mg/ m2 * patient's body surface area, d2-d15 was taken orally by Digio, 20mg three times a day each time. Cetuximab combined with chemotherapy was administered intravenously, once every three weeks, before oxaliplatin, and the dosage was 250mg/ m2 * patient's body surface area. Metronidazole 0.4g/ time, once a day; Vitamin A 25,000 units/time, once a day; Folic acid 0.4mg/ time, once a day. The last three drugs were continued until the end of all chemotherapy cycles. The above regimen lasted for 6 to 8 sessions, and enrolled patients were reviewed every 3 months for colorectal cancer-related tumor markers, including MRI and CT imaging. The primary endpoint was radiographically confirmed metachronous liver metastases, and the secondary endpoint was death, observed for 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-80 at the time of signing the informed consent;
2. Histologically or cytologically confirmed adenocarcinoma of the colon or rectum;
3. Radical surgery has been performed;
4. Imaging examination showed no liver metastasis;
5. Prehepatic CTC number ≥1;
6. The ECOG performance status is 0-1.
7. No combination of other life-threatening diseases;
8. Willingness and ability to follow scheduled visits, treatment plans, laboratory tests and other research procedures.

Exclusion Criteria:

1. Patients with non-primary colorectal cancer;
2. Patients with liver metastasis or other organ metastasis;
3. Patients without prehepatic CTC or whose prehepatic CTC were negative;
4. People who are severely allergic to one or more of the drugs required in the test;
5. Patients with severe underlying diseases of respiratory, circulatory, urinary and hematopoietic systems.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Metachronous liver metastasis rate | Up to approximately 3 years
  The Metachronous liver metastasis rate is the proportion of CTC-positive patients with metachronous liver metastases after conventional therapy or quintuple method intervention.
Overall Survival (OS) | Up to approximately 3 years
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up. For subjects who survived or were lost to follow-up by the data analysis cutoff date, survival was truncated by the subject's last known survival time.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Zhongguo, Doctor, Study Director — Liaoning Tumor Hospital & Institute Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No